CLINICAL TRIAL: NCT02612519
Title: Alfapump System Versus Transjugular Intrahepatic Portosystemic Shunt and Paracentesis in the Treatment of Ascites. A Multicentre Randomised Controlled Study
Brief Title: Alfapump System Versus Transjugular Intrahepatic Portosystemic Shunt and Paracentesis in the Treatment of Ascites
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitement rate
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Cornelius Engelmann, Dr. med., University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Agua-Trial
Record Dates: First submitted 2015-11-11; First posted 2015-11-23 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Alfapump - Substudy 1 (Experimental): Alfapump implantation
  Interventions: Device: Alfapump
- TIPS - Substudy 1 (Active Comparator): TIPS implantation
  Interventions: Device: TIPS
- Alfapump - Substudy 2 (Experimental): Alfapump implantation
  Interventions: Device: Alfapump
- Standard - Substudy 2 (No Intervention): Standard treatment

INTERVENTIONS:
Device: Alfapump — Implantation of Alfapump
  Arms: Alfapump - Substudy 1; Alfapump - Substudy 2
Device: TIPS — Implantation of TIPS
  Arms: TIPS - Substudy 1

SUMMARY:
Multicentre, open, randomised, and controlled trial conducted in patients diagnosed with recurrent/refractory ascites who meet inclusion/exclusion criteria. The efficacy of the Alfapump, TIPS and paracentesis with regard to the treatment of ascites will be compared. All patients will receive medical care for cirrhosis and ascites according to the institution's standards of care. Standard of care may include, but is not limited to the administration of diuretics, paracentesis and consideration for orthotopic liver transplantation.

DETAILED DESCRIPTION:
The study will include patients with decompensated liver cirrhosis and recurrent or refractory, with regular requirements for large volume paracentesis (see subject inclusion criteria). With respect to TIPS-contraindications patients will be assigned to two substudies. If no TIPS-contraindications exists (sub-study 1) patients will be randomized to Alfapump or TIPS. The presence of at least one TIPS-contraindication (sub-study 2) is leading to a randomization to Alfapump or standard of care. All patients will receive medical care for cirrhosis and ascites according to the institution's standards medical care. Standard of care may include, but is not limited to, administration of diuretics, paracentesis and consideration for orthotopic liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis of the liver
2. Recurrent or refractory ascites
3. Age ≥ 18 years (at informed consent)
4. Written informed consent
5. Expected ability to operate the Alfapump device
6. Alcohol abstinence ≥ 3 months at date of inclusion

Exclusion Criteria:

1. General contraindications indicating an advanced stage of liver cirrhosis:

   * Bilirubin > 5 mg/dl and/or
   * INR > 1.5 (without oral anticoagulant such as Vitamin K antagonists or new oral anticoagulants (NOAKs), which inhibit the determination of INR. Therefore patients must be switched to alternative anticoagulants such as heparin or low molecular heparin or fondaparinux that do not interfere with INR measurements) and/or
   * Serum-Sodium < 130 mmol/l and/or
   * ECOG > 2 (Performance status)
2. Gastrointestinal haemorrhage during the last 7 days before inclusion
3. Renal failure defined as serum creatinine higher than or equal to 1,5 mg/dl at time of inclusion
4. Clinical evidence of recurring bacterial peritonitis, defined as 2 or more episodes over the last 6 months or a single episode within the last 2 weeks before inclusion.
5. Clinical evidence of recurring urinary infections, defined as 2 or more episodes over the last 6 months or a single episode within the last 2 weeks before inclusion.
6. Clinical evidence of loculated ascites.
7. Residual urinary volume exceeding 100 ml if obstructive uropathy is known or suspected
8. Known bladder anomaly which might contraindicate implantation of the device.
9. Known or suspected hepatic or extra hepatic malignancy, unless adequately treated and in complete remission for ≥ 3 years
10. Known active chronic hepatitis C (unless adequately treated, i.e no Virus-RNA detectable after cessation of antiviral treatment)
11. Acute peritonitis
12. Pregnant or nursing women. (A serum pregnancy test is required for fertile women within two years of their last menstruation.)
13. Fertile women (within two years of their last menstruation) without appropriate contraceptive measures (implantation, injections, oral contraceptives, intrauterine devices, partner with vasectomy) while participating in the trial
14. Suspected lack of compliance
15. Patients enrolled in another interventional clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-11; Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the (average) number of paracenteses per quarter during time without device abandonment, transplant, or death documented on a time horizon of 4 quarters (i.e.1 year). | Starts with randomisation and ends after 12 months or when a device abandonment, transplant, or death occurs before.

SECONDARY OUTCOMES:
Number of paracenteses per quarter during time without device abandonment, transplant, or death documented on a time horizon of 24 months. | Starts with randomisation and ends after 24 months or when a device abandonment, transplant, or death occurs before.
Number of paracenteses per quarter during time without transplant or death documented on a time horizon of 24 months. | Starts with randomisation and ends after 24 months or when transplant or death occurs before.
Transplant-free survival | From randomisation to 24 months or to death, censoring patients alive at the date of last information or at the date of orthotopic liver transplantation.
Cumulative Incidence of device abandonment | Starts with randomisation and ends after 24 months or when transplant or death occurs before.
Volume of ascites removed | Starting four weeks after study inclusion and ending after 24 months or when transplant or death occurs before.
Patients Quality of Life (EQ-5D Questionnaire) | Starts with randomisation and ends after 24 months or when transplant or death occurs before.
Frequency and duration of hospital stays | Starts with randomisation and ends after 24 months or when transplant or death occurs before.
Nutrition status, assessed by time course of upper arm girth [cm] | Starts with randomisation and ends after 24 months or when transplant or death occurs before.
Albumin substitution, assessed as total amount per quarter [g]. | Starts with randomisation and ends after 24 months or when transplant or death occurs before.
Cumulative incidence of first occurrence of hepatic encephalopathy Stage 2 or higher | Starts with randomisation and ends after 12 months months or when a device abandonment, transplant, or death occurs before.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Berg, Prof. Dr., Principal Investigator — Uniklinik Leipzig Sektion Hepatologie
Locations (3):
- Germany (3):
  - Medizische Klinik III, Aachen
  - Medizinische Klinik und Poliklinik 1 - Gastroenterologie, Dresden
  - Uniklinik Leipzig, Leipzig